CLINICAL TRIAL: NCT07069868
Title: Telehealth as a Nursing Strategy for Monitoring Patients in an Ambulatory Oncology Phase I Clinical Trial Unit
Brief Title: Telehealth in an Ambulatory Oncology Phase I Clinical Trial Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Deborah M. Melonas, R.N, Registered Nurse, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021P001318
Record Dates: First submitted 2025-01-24; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2021-06

CONDITIONS: Malignant Neoplasm
Keywords: telemedicine; nursing; Phase 1 oncology clinical trial
MeSH Terms: conditions — Neoplasms | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: A quasi-experimental study of weekly telehealth visits was conducted using a single-group repeated measures design for adults with cancer enrolled in cycle one Phase 1 clinical trials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Telehealth visit (Experimental): Patients were approached to participate in up to four nursing telehealth visits during their cycle one Phase 1 oncology clinical trial. Nursing assessed for potential adverse events and dose limiting toxicities using the Common Terminology Criteria for Adverse Events. Previous education was reinforced for participants. If the participant was administering an oral study medication at home, dosing instructions were reviewed, and diary evaluated for proper administration and documentation.
  Interventions: Other: Telehealth

INTERVENTIONS:
Other: Telehealth — During cycle one, participants will be asked about fevers, mucositis, nausea, vomiting, constipation, diarrhea, dyspnea, cough, rash, pain and fever. Symptoms will be graded according to Common Terminology Criteria for Adverse Events. A new adverse event of grade one or higher will be reported to a provider. An adverse event grade two or higher above baseline and/or experiencing cancer related symptoms above baseline, the findings will be reported to a Provider.
  Other Names: Telemedicine

SUMMARY:
The study aimed to evaluate the feasibility, acceptability, satisfaction and effectiveness of telehealth on early identification and mitigation of adverse events during cycle one of a Phase 1 oncology clinical trial.

DETAILED DESCRIPTION:
Oncology patients in Phase 1 clinical trials receive study medications administered for the first time in humans. Participants need to be monitored closely for adverse events which can be serious and have critical implications.

A single group repeated measures design was used to evaluate the effect of telehealth on patient outcomes and patient experience for up to four telehealth sessions and nursing staff perceptions of telehealth. Enrollment was limited to 21 participants, in order to limit the number of patients for a pilot study.

Telehealth sessions began within seven days after the initial treatment and occurred weekly during cycle one of the participant's Phase 1 protocol. Side effects assessed by nursing included mucositis, nausea, vomiting, constipation, diarrhea, dyspnea, cough, rash, pain and fever. Patients were also given the opportunity to address other symptoms.

Original research was required to establish validity of telehealth for managing adverse events, dose limiting toxicities of study medications, and enhancing safe clinical care with potentially meeting unmet patient needs when beginning an oncology Phase 1 clinical trial.

Data Collection tools included:

1. Data collection Table which includes variables, sources of data and timeframes
2. Charlson Comorbidity Index (CCI)
3. Patient Reported Outcomes-Common Terminology for Adverse Events (PRO-CTCAE)
4. Adverse Event for Mucositis
5. Adverse Event for Nausea
6. Adverse Event for Vomiting
7. Adverse Event for Constipation
8. Adverse Event for Diarrhea
9. Adverse Event for Dyspnea
10. Adverse Event for Cough
11. Adverse Event for Acneiform Rash
12. Adverse Event for Maculo-Papular Rash
13. Adverse Event for Pain
14. Adverse Event for Fever
15. Nursing Perception of Telehealth Survey
16. Feasibility of Intervention Measure (FIM). Nursing Perspective on the Feasibility of Utilizing Telehealth Technology Survey
17. Nursing Experience with Telehealth and Patients' Adverse Events Survey
18. Patient Feasibility Survey
19. Acceptability of Intervention Measure (AIM). Patient Experience with Accessibility Related to Telehealth Sessions
20. Patient Experience with Telehealth Survey

ELIGIBILITY:
Inclusion Criteria:

* Cancer diagnosis
* Consented and registered to a Phase I oncology clinical trial
* Cycle one patient
* 18 years of age or older
* Willing to participate in weekly telehealth sessions during cycle one
* Patient Gateway account
* Zoom video application downloaded and installed
* A reliable internet connection
* A device with the following requirements

PC/Mac with:

1. Chrome or Firefox as an internet browser
2. Webcam
3. Microphone
4. Speakers or Headphones

iPhone/iPad/Android Device with:

1. The Partners Patient Gateway Application
2. Front facing camera

Exclusion Criteria:

* Adults who are unable to consent
* Individuals younger than 18 years old
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
The study will be feasible as measured by the Feasibility of Intervention at study completion. | From enrollment to the end of cycle one which can be up to 28 days.
  Measures were scored via a Linkert scale ranging from 1 to 5. The higher the score indicates feasibility. 1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree and 5 = completely agree. Feasibility was measured by patients and nurses to see if telehealth would be feasible if implemented in a Phase 1 oncology clinical trial unit.

SECONDARY OUTCOMES:
The study will be acceptable as measured by the Acceptability of Intervention Measure at study completion. | From enrollment to the end of cycle one which can be up to 28 days.
  Measures were scored via a Linkert scale ranging from 1 to 5. The higher the score indicates acceptability. 1 = completely disagree, 2 = disagree, 3 = neither agree nor disagree, 4 = agree and 5 = completely agree. Acceptability was measured by patients and nurses to see if telehealth would be acceptable for patients and staff in a Phase 1 oncology clinical trial unit.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Melonas, RN, OCN, ASN, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No